CLINICAL TRIAL: NCT02365285
Title: Racial Differences in Vagal Control of Glucose Homeostasis
Acronym: RDVCGH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Principal Investigator, Cyndya Shibao, Medical Doctor, Assistant Professor of Medicine, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 141552
Record Dates: First submitted 2015-01-28; First posted 2015-02-18 (Estimated); Results first posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Galantamine; soybean oil, phospholipid emulsion; Heparin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Galantamine 16 mg then placebo (Experimental): Galantamine 16 mg po one time dose then placebo on 2nd visit
  Interventions: Drug: Galantamine; Drug: Placebo Oral Capsule; Drug: Intralipid; Drug: Heparin
- Placebo then Galantamine 16 mg (Placebo Comparator): Placebo capsule po one time dose then Galantamine 16 mg on 2nd visit
  Interventions: Drug: Galantamine; Drug: Placebo Oral Capsule; Drug: Intralipid; Drug: Heparin

INTERVENTIONS:
Drug: Galantamine — 16 mg po prior to the infusion of intralipid
  Other Names: Razadyne
Drug: Placebo Oral Capsule — Placebo oral capsule prior to the infusion of intralipid/heparin
Drug: Intralipid — Intralipid 20% will be infused at 0.8 mL/m2/min for 4h after oral placebo or Galantamine
  Other Names: I.V. Fat Emulsion
Drug: Heparin — heparin bolus of 1000 U will be followed by 200 U/h infusion for 4h after oral placebo or Galantamine

SUMMARY:
The investigators will test the hypothesis that acute central acetylcholinesterase inhibition will restore PNS activity and reduce oxidation in AAW compared to whites.

DETAILED DESCRIPTION:
Obesity has a greater detrimental impact on the health of African American women (AAW) than on any other racial or gender group. Nearly 80% of AAW are overweight or obese. Reduced insulin sensitivity is more prevalent among AAW as compared to white women and men of both races. This condition puts AAW at increased risk for the development of type 2 diabetes mellitus. The exact mechanism underlying these pathophysiological differences remains unknown. The investigators have found that obese AAW have decreased parasympathetic nerve (PNS) activity compared to whites and recent studies in animal models showed that the PNS confers protection against oxidative stress. In our AA cohort, PNS activity was directly correlated with insulin sensitivity in obese AAW even after controlling for differences in age, blood pressure and visceral adiposity. Equally important, the investigators also showed that the decrease in insulin sensitivity was associated with increased oxidative stress as measured by plasma levels of F2-isoprostanes. Taken together these findings lead us to hypothesize that the decreased PNS activity in obese AAW compared to white women has deleterious effects on oxidative stress and insulin sensitivity.The investigators will test the hypothesis that acute central acetylcholinesterase inhibition will restore PNS activity and reduce oxidation in AAW compared to whites.

ELIGIBILITY:
Inclusion Criteria:

* Female
* African American or white (race will be self-defined, but only subjects who report both parents of the same race will be included)
* 18-60 years old
* BMI 30-45 Kg/m2
* Not pregnant or breastfeeding

Exclusion Criteria:

* Pregnant or breastfeeding
* Diabetes diagnosis (defined by the American Diabetes Association (ADA) criteria)38
* Cardiovascular disease such as myocardial infarction within 6 months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, mitral valve stenosis, aortic stenosis, or hypertrophic cardiomyopathy.
* Arrhythmia (first-, second-, and third-degree atrioventricular (AV) block)
* Significant weight change >5% in the past 3 months
* Impaired hepatic function (AST and/or Alanine transaminase (ALT) > one and one half times (1.5X) upper limit of normal range)
* Impaired renal function (eGFR <60ml/min)
* Users of strong inhibitors of Cytochrome P450 3A4 (CYP3A4) or cytochrome P450, family 2, subfamily D, polypeptide 6 (CYP2D6)
* Users of other acetylcholinesterase inhibitors such as pyridostigmine or bethanechol
* History of alcohol or drug abuse
* Mental conditions rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Inability to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cyndya Shibao, MD, Principal Investigator — Vanderbilt University Medical Center, Clinical Pharmacology
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Parsa D, Aden LA, Pitzer A, Ding T, Yu C, Diedrich A, Milne GL, Kirabo A, Shibao CA. Enhanced parasympathetic cholinergic activity with galantamine inhibited lipid-induced oxidative stress in obese African Americans. Mol Med. 2022 Jun 3;28(1):60. doi: 10.1186/s10020-022-00486-5. PMID 35659521

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 52 participants were screen failures and did not receive an intervention.
Groups:
- Galantamine 16 mg Then Placebo (African-American); Galantamine 16 mg Then Placebo (White): Galantamine 16 mg po one time dose then placebo on 2nd visit
  Intralipid: Intralipid 20% will be infused at 0.8 mL/m2/min for 4h after oral placebo or Galantamine
  Heparin: heparin bolus of 1000 U will be followed by 200 U/h infusion for 4h after oral placebo or Galantamine
- Placebo Then Galantamine 16 mg (African-American); Placebo Then Galantamine 16 mg (White): Placebo capsule po one time dose then Galantamine 16 mg on 2nd visit
  Intralipid: Intralipid 20% will be infused at 0.8 mL/m2/min for 4h after oral placebo or Galantamine
  Heparin: heparin bolus of 1000 U will be followed by 200 U/h infusion for 4h after oral placebo or Galantamine
Period: Overall Study
Arm/Group | Galantamine 16 mg Then Placebo (African-American) | Galantamine 16 mg Then Placebo (White) | Placebo Then Galantamine 16 mg (African-American) | Placebo Then Galantamine 16 mg (White)
Started | 7 | 6 | 7 | 3
Completed | 7 | 5 | 6 | 1
Not Completed | 0 | 1 | 1 | 2
Not completed — Physician Decision | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Galantamine 16 mg Then Placebo (African-American) | Galantamine 16 mg Then Placebo (White) | Placebo Then Galantamine 16 mg (African-American) | Placebo Then Galantamine 16 mg (White) | Total
Number analyzed (Participants) | 7 | 6 | 7 | 3 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 7 | 3 | 23
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 7 | 3 | 23
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 0 | 7 | 0 | 14
  White | 0 | 6 | 0 | 3 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 7 | 3 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Oxidative Stress: Baseline to 2 Hours
Description: Measure F-2 isoprostanes as a marker of oxidation
Time Frame: Baseline to 2 hours
Population: 2 white participants dropped out due to nausea. 1 African-American was withdrawn, MD decision.
Measure: Mean (Standard Deviation); unit: pg /ml
Groups:
- Galantamine 16 mg (African-American); Galantamine 16 mg (White): Galantamine 16 mg po one time dose
  Intralipid: Intralipid 20% will be infused at 0.8 mL/m2/min for 4h after oral placebo or Galantamine
  Heparin: heparin bolus of 1000 U will be followed by 200 U/h infusion for 4h after oral placebo or Galantamine
- Placebo (African-American); Placebo (White): Placebo capsule po one time dose
  Intralipid: Intralipid 20% will be infused at 0.8 mL/m2/min for 4h after oral placebo or Galantamine
  Heparin: heparin bolus of 1000 U will be followed by 200 U/h infusion for 4h after oral placebo or Galantamine
Arm/Group | Galantamine 16 mg (African-American) | Galantamine 16 mg (White) | Placebo (African-American) | Placebo (White)
Number analyzed (Participants) | 13 | 7 | 13 | 7
pg /ml | -0.003 (0.012) | -0.006 (0.018) | 0.01 (0.018) | -0.006 (0.01)

2. Primary Outcome: Change in Oxidative Stress: Baseline to 4 Hours
Description: Measure F-2 isoprostanes as a marker of oxidation
Time Frame: Baseline to 4 hours
Population: 1 white participant did not have 4 hour F-2 isoprostanes drawn after receiving placebo. 2 white participants dropped out due to nausea. 1 African-American was withdrawn, MD decision.
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Galantamine 16 mg(White): Galantamine 16 mg po one time dose
  Intralipid: Intralipid 20% will be infused at 0.8 mL/m2/min for 4h after oral placebo or Galantamine
  Heparin: heparin bolus of 1000 U will be followed by 200 U/h infusion for 4h after oral placebo or Galantamine
- Placebo(White): Placebo capsule po one time dose
  Intralipid: Intralipid 20% will be infused at 0.8 mL/m2/min for 4h after oral placebo or Galantamine
  Heparin: heparin bolus of 1000 U will be followed by 200 U/h infusion for 4h after oral placebo or Galantamine
Arm/Group | Galantamine 16 mg (African-American) | Galantamine 16 mg(White) | Placebo (African-American) | Placebo(White)
Number analyzed (Participants) | 13 | 7 | 13 | 6
pg/ml | 0 (0.016) | -0.008 (0.014) | 0.003 (0.005) | -0.008 (0.014)

ADVERSE EVENTS:
Time Frame: Baseline through 2nd study day, usually about 1 month.
Arm/Group | Galantamine 16 mg (African-American) | Galantamine 16 mg (White) | Placebo (African-American) | Placebo (White)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/9 | 0/14 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/9 | 0/14 | 0/9
Other Adverse Events (participants affected / at risk) | 4/14 | 6/9 | 2/14 | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Galantamine 16 mg (African-American) (N=14) | Galantamine 16 mg (White) (N=9) | Placebo (African-American) (N=14) | Placebo (White) (N=9)
Nausea and Vomiting (Gastrointestinal disorders) | 3 (3) | 5 (5) | 2 (2) | 1 (1)
Lightheadness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT02365285/Prot_SAP_000.pdf